CLINICAL TRIAL: NCT04522505
Title: Long-term Follow-up for Safety Evaluation of Subjects Who Participated in the Phase 1 Clinical Trial of CS20AT04(CS20AT04-LN101) in Lupus Nephritis
Brief Title: Long-term Follow-up for Evaluating the Safety of CS20AT04 in Subject with Lupus Nephritis
Status: Completed | Type: Observational
Sponsor: Corestemchemon, Inc. (Industry)
Collaborators: Hanyang University (Other)
Responsible Party: Sponsor
Other Study IDs: CS20AT04-LN101-E
Record Dates: First submitted 2020-07-01; First posted 2020-08-21 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Lupus Nephritis
Keywords: Systemic lupus erythematosus; Allogenic bone marrow derived mesenchymal stem cell
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This observation study is planned to evaluate the safety and efficacy of the subjects who received CS20AT04 in the phase 1 clinical trial.

If the subjects who participated in the phase 1 clinical trial voluntarily agree to participate in this observation study, visit 1 and visit 2 will be conducted every 3 months according to the clinical trial protocol until 6 months after administration of CS20AT04 in the phase 1 clinical trial. And Visit 3 after 6 months, Visit 4~Visit 7 will be conducted every 12 months. During each visit, subjects are assessed for the efficacy and occurrence of adverse events.

DETAILED DESCRIPTION:
Lupus is a representative autoimmune disease that affects the whole body. It is occurred by generation of autoantibody and immune complex due to abnormal activation of the immune cells on the basis of abnormal immune responses.

Although about 50% of lupus patients have lupus nephritis, there is no therapeutic product targeting for the lupus nephritis so far.

The investigator has performed the pre-clinical and clinical studies using allogenic bone marrow derived mesenchymal stem cells in SLE.

CS20AT04 has anti-inflammatory effects, controls activity of immune cells and reduces generation of autoantibodies. So, it is expected to have therapeutic effects on lupus nephritis.

Phase 1 clinical trial was conducted as a single center, open-label.

The main component of CS20AT04 is bone marrow-derived mesenchymal stem cells. And the risk of tumor formation is low. Through the repeated administration and long-term observation with mouse model, it was confirmed that there was no oncogenicity. In addition, it was confirmed through the cell residual tracking test of the animal model that the in vivo residual period was shorter than 14 days.

However, since long-term safety has not been evaluated after administering CS20AT04 to humans, the investigator will confirm the safety of stem cells for up to 5 years according to the risk management plan for stem cell products of the Ministry of Food and Drug Safety and already approved phase 1 clinical trial.

Also In the phase 1 clinical trial that only confirmed safety and tolerability for 28 days after administration of CS20AT04, it is difficult to confirm the continuous change of the indicator for evaluating efficacy.

So, it is necessary to check the efficacy in this observation study.

ELIGIBILITY:
Inclusion Criteria:

* A Person who enrolled in a phase 1 clinical trial using CS20AT04 (CS20AT04-LN101) and administered CS20AT04 and has been 3 months.
* A person who voluntarily consent to participate in this observational study

  *Phase I clinical trial Inclusion Criteria
* Patients with HLA-haplo-matched bone marrow donor is less than 70 years old.
* Clinical diagnosis of SLE by American College of Rheumatology (ACR) criteria.
* Patients had suffered from active renal disease in the past or patients has active renal disease now. Active renal disese should have include below.

Spot urine protein/creatinine ratio ≥ 1.0 and ① >5 RBC/HPF, ② >5 WBC/HPF, ③ columnar cell.

Biopsy confirmed active type III or type IV, or type V lupus nephritis. Patients can be immunosuppressive agent to , steroids, taking, such as anti-Malarials (hydroxychloroquine) in a certain capacity, during the test period, to maintain the same capacity before 4-weeks screening.

Patients who consented to participate in the study in writing by themselves or their legal representatives.

Exclusion Criteria:

* A person who do not agree to participate in this follow up observational study among the subjects enrolled in a phase 1 clinical trial using CS20AT04.

  *Phase I clinical trial exclusion criteria
* Those who do not kidney disease for SLE.
* Patients with a history of hypersensitivity, such as heavy metal poisoning similar to drug testing and drug ingredients.
* Patients a history Major organs (kidney, liver, lung, heart) transplant or liver hematopoietic cells / transplant or during of scheduled transplantation clinical trial.
* patients a history of kidney dialysis or during of the scheduled dialysis clinical trials within 2 weeks prior to the screening.
* Tested positive for hepatitis B(HBsAg, Anti-HBcAB, HBV-DNA) and hepatitis C(Anti-HCV, HCV-RNA).
* Patients a history of anaphylactic reaction for the parenteral administration of a monoclonal antibody or contrast agent, a mouse protein or human.
* Patients whose e-GFR ≤ 30mL/min at screening.
* Patients with a history of malignancy within 5 years prior to the screening(basal cell carcinoma of skin, squamous cell carcinoma of skin, or cervical intraepithelial neoplasia are excluded).
* Patients who were administered drug of the follow within 6 months prior to the screening.

nitrogen mustard, chlorambucil, vin·cris·tine, procarbazine, Abatacept, Rituximab, Belimumab Patients who were administered drug of the follow within 3 months prior to the screening.

Anti-TNF therapy(Etanercept, adalimumab, Infliximab, golimumab, Tocilizumab) Interleukin-1 receptor antagonist(anakinra) Intravenous immunoglobulin(IVIG) Plasmapheresis

* Those who are hypersensitive to antibiotics including penicillin and streptomycin.
* Patients with systemic infection at screening.
* Uncontrolled hypertension or diabetes.
* If that may affect proteinuria increased capacity or begin taking medication(ACE inhibitors, ARB (Angiotensin Receptor Blocker)) (However, more than four weeks allowed capacity, taking is possible during the trial period without changing capacity).
* Patients who showed myocardial infarction or angina on ECG at screening, or received stent procedure or bypass.
* Patients who were administered another study drug 3 months prior to the study.
* Patients with severe mental disease(for example, schizophrenia, bipolar disorder etc;).
* Patients are expected to be administered the combination contraindicated drugs about inevitable or taker within clinical trial.
* Women of childbearing age are not implement adequate contraception during clinical trials. the proper method of contraception, which has Oral contraceptive continued more than four weeks, a surgical procedures including the insertion loop, condom use etc. and Medically it is determined that there is no possibility of pregnant women do not belong to women of childbearing age due to the ovary removal, hysterectomy and menopause, etc.
* Pregnant women or nursing women.
* Except as permitted in the following Case and laboratory test results than moderate adverse events(NCI-CTC (National Cancer Institute-Common Toxicity Criteria) version 4.0) grade 3.
* Class III due to stable prothrombin time of warfarin therapy
* Lupus anticoagulant group, and are not associated with liver disease or stable anticoagulation 3 grade partial thromboplastin time
* Lupus due to hepatitis and alcoholic liver disease, are not associated with uncontrolled diabetes or viral hepatitis stable 3 grade gamma glutamyl transferase (GGT) increases. If it appears to be less than ALT and / or AST is above all on the second level.
* Stable grade 3 neutropenia or white blood cell count
* Patients who previously received stem cell therapy.
* Subjects who by the investigator to make them ineligible for participation in this clinical study.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Patients with HLA-haplo-matched bone marrow donor is less than 70 years old.
  * Clinical diagnosis of SLE by American College of Rheumatology (ACR) criteria.
  * Patients had suffered from active renal disease in the past or patients has active renal disease now.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | up to 57 months after enrollment
  After the completion of the CS20AT04-LN101 phase 1 trail, new adverse events, including tumor are assessed and detailed information is collected at each visit.
Incidence of abnormal results of Physical examination | up to 57 months after enrollment
  Physical examination is performed at each visit. If clinically significant abnormal findings are recorded in the CRF and collected as AEs.
Percentage of abnormal Vital signs | up to 57 months after enrollment
  Percentage of abnormal Blood pressure (mmHg) and Pulse rate (beat per minute)
Percentage of abnormal results of Laboratory tests | up to 57 months after enrollment
  The following laboratory tests are performed at each visit
  * Hematology test: WBC, RBC, Hemoglobin, Hematocrit, Platelet count, WBC Diffcount, ESR
  * Chemistry test : Total protein, Albumin, Total bilirubin, SGOT(AST), SGPT(ALT), rGTP, Sodium, Potassium, BUN, Creatinine, Glucose, Alkaline Phosphatase, Chloride, Total cholesterol, Triglyceride, Uric Acid , CPK, LDH, CRP, Adolase
  * Urine analysis : Protein, Creatinine, Glucose, Urobilinogen, WBC, RBC, Urine Sediment, Creatinine, Urine albumin creatinine ratio, Urine protein creatinine ratio

SECONDARY OUTCOMES:
SLEDAI-2K (Systemic Lupus Erythematosus Disease Activity Index-2000) | up to 57 months after enrollment
  Evaluate disease activity of 9 organ systems and display it as a score. The score is weighted from 1 to 8 at each system, if descriptor is present at the time of visit or in the proceeding 10 days.
  * Change in SLEDAI>3 points means mild or moderate flare
  * Change in SLEDAI>12 points means severe flare
BILAG 2004 (British Isles Lupus Assessment Group 2004) | up to 57 months after enrollment
  The change in disease activity in the last 4 weeks compared to the previous 4 weeks is evaluated as score.
SDI (Systemic Lupus International Collaborating Clinics/Americans College of Rheumatology (SLICC/ACR) Damage Index | up to 57 months after enrollment
  Only if the damage due to the disease lasted for at least 6 months is evaluated on a scale 0-47.
Disease activity assessed by PGA (Physician Global Assessment) | up to 57 months after enrollment
  Investigator evaluated disease activity in mm using 0 to 100mm visual analogue scale (VAS). High score indicates worsening of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: SANG-CHEOL BAE, M.D.,Ph.D., Principal Investigator — Hanyang University
Locations (1):
- Hanyang university hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided